CLINICAL TRIAL: NCT01649596
Title: Impact of Expanded Peri Operative Warming for Patients Undergoing Elective Surgery
Brief Title: Impact of Expanded Peri Operative Warming
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension Health (Industry)
Collaborators: 3M (Industry)
Responsible Party: Principal Investigator, Tarik Wasfie, MD, MD, General Surgeon, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GRMC120009
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Hypothermia; Complications
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Masking Description: Open label.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warming Gown (Active Comparator): Comparison of two types of warming processes prior to, during, and after the surgery procedure.
  Interventions: Device: Warming Gown
- Standard of Care Warming (Other): Standard of care warming with hospital-issued blankets.
  Interventions: Other: Standard of care warming

INTERVENTIONS:
Device: Warming Gown — Forced air warming Gown and portable warming unit that follows patient from pre-operative through surgery and into post-operative recovery.
  Other Names: 3M Bair Paws Flex Gown and Bair Paws Model 875 Warmer
  Arms: Warming Gown
Other: Standard of care warming — The intervention is standard of care, placing warm blankets on the patient at time of pre operative preparation through the procedure and into recovery.
  Arms: Standard of Care Warming

SUMMARY:
The purpose of this proposed study is to evaluate a normothermia protocol that includes preoperative warming and standard intra operative temperature management in patients undergoing general surgery.

DETAILED DESCRIPTION:
This study was designed to evaluate a normothermia protocol that includes preoperative warming and standard intra operative temperature management in patients undergoing general surgery. It compares short term outcomes in patients for whom warming is expanded by commencing in the pre operative area and is maintained through post operative recovery versus patients receiving the standard warming at time of induction. Patients were randomly assigned to either a warming blanket device or standard warming procedures. The study tested for differences in the rate of hypothermic events between the two groups. A secondary goal was to test for differences in the complication rate and patient satisfaction between the two groups.

This study is testing the hypothesis that expanded warming significantly reduces rates of hypothermia and complications over standard warming used only during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are adult patients 18 years and older elective surgery of > 1 hour

Exclusion Criteria:

* Emergency and/or trauma cases
* Patients with diminished mental capacity unable to fill out or respond to survey questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarik Wasfie, MD, Principal Investigator — Ascension Health
Locations (1):
- Genesys Regional Medical Center, Grand Blanc, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual data was de-identified and not available to share on an individual level. Aggregate data was planned to shared by publishing in a scientific journal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inpatients having surgery between September 1, 2012 through April 9, 2013.
Pre-assignment Details: Patients presenting with emergencies or with trauma were excluded.
Groups:
- 3M Bair Paws Flex Gown: 3M Bair Paws Flex Warming Gown and 3M Bair Paws Model 875 Warming Unit
  3M Bair Paws Flex Gown and Bair Paws Model 875 Warmer
- Control: Standard of care warm blankets
Period: Overall Study
Arm/Group | 3M Bair Paws Flex Gown | Control
Started | 46 | 48
Completed | 46 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 94 subjects were included. Average age was 50.1 years. Overall, 69% were female and 90% were Caucasian. The mean core temperature in pre-op for the extended warming group was 36.8 degrees and for the control group was 36.6 degrees.
Groups:
- Control: Standard of care, warm blankets
  Standard of care - warm blankets
- Total: Total of all reporting groups
Arm/Group | 3M Bair Paws Flex Gown | Control | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (14.9) | 48.5 (15.1) | 50.1 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 28 | 65
  Male | 9 | 20 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 41 | 44 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94
BMI [Mean (Standard Deviation); unit: Kg/m^2] | 32.6 (7.9) | 29.8 (7.1) | 31.2 (7.6)
Pulse [Mean (Standard Deviation); unit: bpm] | 76.2 (12.2) | 74.2 (15.2) | 75.2 (13.8)
Temperature [Mean (Standard Deviation); unit: Celsius] | 36.8 (0.4) | 36.5 (0.3) | 36.7 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypothermic Events
Description: The primary outcome is the incidence of hypothermic events (core <36 degrees celsius).
Time Frame: 12 hours
Measure: Number; unit: participants
Arm/Group | 3M Bair Paws Flex Gown | Control
Number analyzed (Participants) | 46 | 48
participants | 5 | 10
Statistical Analysis 1: Comparison: 3M Bair Paws Flex Gown vs Control; Test type: Superiority or Other; p = 0.12, Chi-squared; percent = 10

2. Secondary Outcome: Patient Satisfaction
Description: Secondary outcome is the relative change (%) in patient satisfaction score from pre-op to recovery. Pre-procedure and Post-procedure surveys were given to the participants to complete. Pre-procedure survey contained 9 questions and the post-procedure survey contained 6 questions. The questions were related to comfort, anxiety and satisfaction. A questionnaire was designed with 6 questions (2 pt and 4 pt Likert sub scales) combined. The overall scores were additive and ranged from 5 to 18 points (5 indicating the least anxiety and 18 indicating the highest anxiety). Individual scores were summed, averaged and group averages compared. The relative change in the percent of participants satisfied (somewhat & highly) was calculated for each group. The change in percent satisfied was calculated for each group and compared.
Time Frame: 12 hours
Population: All patients completed the patient anxiety and satisfaction survey.
Measure: Number; unit: change in percent satisfied
Arm/Group | 3M Bair Paws Flex Gown | Control
Number analyzed (Participants) | 46 | 48
change in percent satisfied | 59 | 49
Statistical Analysis 1: Comparison: 3M Bair Paws Flex Gown vs Control; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; A t-test for percents was used to compare the number of participants (%) from each group reporting satisfaction (somewhat and highly satisfied); percent = 48

ADVERSE EVENTS:
Arm/Group | 3M Bair Paws Flex Gown | Control
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No